CLINICAL TRIAL: NCT03508479
Title: Study of Airway Inflammatory Responses to Experimental Rhinovirus Infection
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Suspended due to COVID-19. Protocol did not resume post COVID due to funding.
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16-3283
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers; Rhinovirus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RG-HRV16 Inoculation (Experimental): While wearing a dental bib, subjects will be asked to blow the nose prior to inoculation. With the head tilted back, a total of 0.5 mL (0.25 mL/nostril) will be administered using the MAD Nasal™ Intranasal Mucosal Atomization Device. Subjects instructed not to blow nose for 30 minutes afterwards.
  Interventions: Biological: RG-HRV16

INTERVENTIONS:
Biological: RG-HRV16 — 0.25 mL inoculum intranasally delivered into each nostril (0.5 mL total delivered). Total cumulative dose of 1000 median tissue culture infective dose at 50% of cells inoculated (TCID50).
  Other Names: Rhinovirus Type 16

SUMMARY:
This study is designed to characterize in detail the clinical, physiologic, and inflammatory features of Human Rhinovirus (HRV) infection in healthy volunteers without underlying lung disease while also evaluating the safety of HRV administrations.

DETAILED DESCRIPTION:
The majority of severe exacerbations of asthma and need for hospitalizations are triggered by infection with respiratory viruses. Of these, rhinovirus is the most commonly implicated virus. Furthermore, there is evidence that viral infections exert synergistic effects with other stimuli to provoke asthma symptoms such as exposure to allergens and air pollutants. Experimental HRV infection studies have yielded important insights into the underlying disease mechanisms of viral-induced asthma exacerbations, and have been integral to identifying candidates for the development of new therapies. These studies have been safely conducted in both healthy and susceptible populations (those with underlying airway disease such as asthma and chronic obstructive pulmonary disease (COPD)), for more than 60 years.

Much of the understanding of the clinical course of HRV infection is derived from experimental infections of healthy human volunteers. In these studies, subjects were inoculated intranasally with up to 10,000 [tissue culture infectious dose (TCID)] TCID50 of HRV, the most commonly used strains being HRV-16 and HRV-39. Experimental HRV infection produces the hallmark clinical features of the common cold including rhinorrhea and nasal obstruction. Respiratory symptoms typically develop 1-2 days after inoculation. Cold symptom scores generally peak 2-4 days post infection and return to baseline within 1 week in most infected subjects. HRV infection induces changes in inflammatory cell recruitment, nasal cytokine levels, and gene expression, which occur concurrently with clinical symptoms.

While the symptoms of HRV infection are typically limited to the upper respiratory tract in healthy subjects, those with underlying airway disease such asthma and COPD are more likely to exhibit an augmented and prolonged response to HRV infection with lower airway involvement. HRV is the leading viral cause of exacerbations of asthma and COPD; therefore, the response of these populations to HRV infection has been the focus of a number of studies. Although most studies in asthmatics have been performed in inhaled corticosteroid-naïve subjects, a recent study performed in subjects whose asthma was well controlled with inhaled corticosteroids demonstrates the safety of experimental HRV infection in this population. This model has also been employed in conjunction with other exposure models such as allergen challenge and pollutant exposure. There are several ongoing and recently completed clinical trials registered with ClinicalTrials.gov that utilize the HRV infection model. Of these, several employ the HRV-16 strain (ClinicalTrials.gov Identifiers: NCT01769573, NCT01466738, NCT01823640, NCT03073837, NCT03296917, NCT01704040, NCT02910401) being used in this study. Both healthy and asthmatic volunteers are represented in these clinical trials.

In summary, the experimental HRV infection model has proven to be a safe and valuable tool for examining various aspects of HRV biology. Due to the limitations associated with animal models of asthma and COPD, and the lack of animal species that are permissive for HRVs, experimental infection of humans with HRV has been integral for examining the pathophysiology of virus-induced exacerbations of asthma and COPD. Although experimental HRV-infection results in a reduction in lung function for some asthmatics and COPD patients, no serious adverse events have been reported using this model.

The goal of this study is to establish the experimental HRV-infection model in this research center using a viral inoculum referred to as RG-HRV-16. This strain was used in a recently-completed safety and dosing study (NCT01769573). Our study would provide the pilot data needed for the design of subsequent studies evaluating innate immune responses to HRV infection in asthmatics, modulation of HRV-induced responses by inhaled pollutants, and efficacy of novel therapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years of either gender
2. Non-smoker (less than 10 cigarettes per month for at least the prior 3 years)
3. Negative pregnancy test (for females as applicable)
4. Oxygen saturation of > 94% and blood pressure with systolic value between 140-90 mm Hg and diastolic between 80-55 mm Hg
5. Willingness to hold all nasal medications (including, but not limited to, nasal steroids or nasal spray decongestants), oral antihistamines and leukotriene inhibitors for at least 1 week prior to Day 0 and continuing throughout the remaining study period.
6. Negative Allergy Skin Test (AST) at a separate screening visit performed prior to study enrollment, University of North Carolina Institutional Review Board (UNC IRB) approved study # 98-0799, Database and Screening Protocol for Research Studies of the Center for Environmental Medicine and Lung Biology (CEMALB). (Results from AST performed within the past 12 months as part of another study protocol or AST reports from testing performed by the subject's Medical Doctor (MD) within the past 12 months will also be accepted.)
7. Negative methacholine inhalation challenge as performed in the separate screening protocol. (Less than a 20% decrease in Forced Exhaled Volume at 1 second (FEV1) at a maximum methacholine concentration of 10 mg/ml).
8. Normal lung function, defined as (NHANES III predicted set):

   * Forced Vital Capacity (FVC) of ≥ 80 % of that predicted for gender, ethnicity, age and height
   * FEV1 of ≥ 80 % of that predicted for gender, ethnicity, age and height
   * Ratio of Forced Exhaled Volume at 1 second to Forced Vital Capacity (FEV1/FVC) ≥ .75
9. No nasal symptoms, based on respiratory questionnaire

Exclusion Criteria:

1. Presence of neutralizing antibodies to RG-HRV-16 at the screening visit to a titer of ≥ 1:2.
2. Inability or unwillingness of a participant to give written informed consent
3. History of rhinitis, chronic sinusitis, or other sinus disease, or any chronic cardiorespiratory disease
4. Subjects with household contacts with chronic lung disease, who are children under the age of 2 years, and who are adults over the age of 65 years
5. Subjects who live in communal settings (i.e. dormitories)
6. Respiratory infection (cough, sore throat, sinusitis, fever etc) within prior 4 weeks
7. Received any live vaccine in the past 4 weeks or an inactivated vaccine within the past 2 weeks
8. Active wheezing at the time of the Day 0 visit
9. Pregnancy or nursing or women who are currently trying to become pregnant; all female subjects, except those who have had a hysterectomy with oophorectomy, will undergo urine pregnancy testing on the morning of the screening visit and again on the on Day 0 at the time of arrival to the lab and prior to HRV administration. A positive pregnancy test will exclude the subject
10. History of any immunosuppressive disease or a positive Human immunodeficiency virus (HIV) test at the screening visit
11. Use of immunosuppressive drugs within the past 6 months
12. Chronic medications which, in the opinion of the study physician(s), may either increase the risks of participation or may interfere with the findings of the study
13. Current use of beta-adrenergic blocking agents
14. Current use of antidepressants if classified as tricyclic or Monoamine oxidase inhibitors (MAO) inhibitors;
15. Known hypersensitivity to methacholine or to other parasympathomimetic agents;
16. History of fainting or feeling severely dizzy with blood draws
17. History of Guillain-Barre syndrome
18. Subjects who will be unable to avoid contact with immunocompromised individuals for 3 weeks after receiving RG-HRV16
19. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study;
20. Unwillingness to use reliable contraception if sexually active (Intrauterine Device (IUD), birth control pills/patch, condoms)
21. Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements
22. Participation in any study using an investigational agent within 30 days of enrollment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in neutrophils/mL in nasal lavage fluid from baseline to mean of days 2-4 post inoculation | Baseline and study visit days 2-4
  Nasal lavage fluid will be collected at baseline. Participants will then undergo RG-HRV16 inoculation. Nasal lavage fluid will be collected on days 2-3 post inoculation and mean neutrophils/ml over days 2-4 will be compared to baseline.

SECONDARY OUTCOMES:
Mean Symptom Score from Cold Symptom Questionnaire up to 4 weeks post-inoculation | 4 weeks post-inoculation
  Assessment of eight clinical symptoms on the day of RG-HRV16 inoculation and days 2, 3, 4, 7, 14, 28 following inoculation will be performed with a cold symptom questionnaire. Scores of 0, 1, 2, or 3 will be given to symptoms rated as absent, mild, moderate, or severe, respectively. Minimum score: 0. Maximum score: 32.
Change in FEV1 and FEF25-75% from baseline to 4 weeks post-inoculation | Baseline and 4 weeks post-inoculation
  Changes in FEV1 and FEF25-75% (mean forced expiratory flow between 25% and 75% of the FVC or maximum mid-expiratory flow) from baseline will be assessed up to 4 weeks post-RG-HRV16 inoculation (on days 2, 3, 4, 7, 14, and 28 following inoculation).
Change in Methacholine reactivity, as measured by the concentration of methacholine resulting in a 20% drop in FEV1 (PC20), from baseline to day 4 post-inoculation | Baseline and study visit day 4 (post-inoculation)
  Participants will undergo a methacholine challenge to assess airway hyper-responsiveness at baseline. Changes in methacholine reactivity, as measured by the PC20, from baseline to 4 days after RG-HRV16 inoculation will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hernandez, MD, Principal Investigator — University of North Carolina
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No